CLINICAL TRIAL: NCT04412369
Title: Multi-modality Imaging & Immunophenotyping of COVID-19 Related Myocardial Injury
Acronym: MIIC-MI
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); British Heart Foundation (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Jason Tarkin, Wellcome Clinical Research Career Development Fellow, University of Cambridge
Other Study IDs: A09565
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: COVID19; Cardiovascular Diseases
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with COVID-19 and cardiac Troponin elevation
  Interventions: Diagnostic Test: Non-invasive cardiac imaging

INTERVENTIONS:
Diagnostic Test: Non-invasive cardiac imaging — Cardiac MRI ± CT coronary angiography ± Cardiac PET/MRI (68Ga-DOTATATE or 18F-FDG)

SUMMARY:
Cardiovascular involvement in coronavirus disease-2019 (COVID-19) encompasses a wide range of vascular and myocardial pathologies, including both acute and long-term sequelae. The MIIC-MI study aims to investigate mechanisms of cardiac injury in COVID-19 using multi-modality imaging and immunophenotyping to better understand the link with adverse patient outcomes.

DETAILED DESCRIPTION:
Cardiovascular involvement in coronavirus disease-2019 (COVID-19) encompasses a wide range of vascular and myocardial pathologies, including both acute and long-term sequelae.

Cardiac Troponin elevation, a marker of acute myocardial injury, has been identified in up to 28% of hospitalized patients with coronavirus disease 2019 (COVID-19) and is associated with an increased mortality risk. However, the predominant aetiology of myocardial injury relating to COVID-19 remains unclear. The Troponin leak could either signify direct cardiac involvement in COVID-19 or serve as a non-specific marker of a severe systemic insult.

There have been numerous reports of acute myocarditis in patients with COVID-19. Other contributory mechanisms of cardiac Troponin elevation in patients with COVID-19 that are also driven by a proinflammatory state include acute myocardial infarction due to atherosclerotic plaque rupture (type 1) or demand ischemia (type 2), endothelial and microvascular dysfunction, immune-mediated activation of coagulation and fibrinolytic systems, and stress cardiomyopathy.

Longer-term effects of COVID-19 on the cardiovascular system are also unknown. Many individuals with post-acute sequalae of SARS-CoV-2 infection (or 'long COVID') have unexplained cardiac symptoms. Patients may also present with new-onset heart failure after COVID-19, which is not attributed to another cause.

We aim to identify patterns of myocardial injury in COVID-19 using non-invasive multi-modality cardiac imaging, paired with cytokine/chemokine testing, immunophenotyping of peripheral blood cells and coagulation profiles.

A better understanding of the mechanisms underlying the excess mortality risk attributable to myocardial injury in COVID-19 is needed and may help to improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Confirmed COVID-19 infection AND Troponin I elevation >99th percentile of upper reference limit OR new-onset heart failure OR unexplained cardiac symptoms
* Able to give written, informed consent

Exclusion Criteria:

* Women of child-bearing potential not using adequate contraception
* Contra-indication to MRI scanning
* Contrast allergy or contrast-nephropathy
* Chronic kidney disease (eGFR <30 mL/min/1.73 m2)
* Previous myocardial infarction
* Uncontrolled atrial fibrillation
* Uncontrolled chronic inflammatory disease
* Severe lymphopenia (<0.2 x109/L)
* Treatment with immunomodulatory therapies within the last month (excluding inhaled or topical steroid therapy)
* Any medical condition, in the opinion of the investigator, that prevents the participant from lying flat during scanning, or from participating in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of COVID-19 and cardiovascular involvement
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis | Baseline
  Number of participants with a diagnosis of COVID-19 related myocarditis, Type 1 or 2 myocardial infarction and/or other mechanism of cardiac injury confirmed by multi-modality imaging.

SECONDARY OUTCOMES:
Immune markers | Baseline
  Comparison of a panel of inflammatory cytokines and immune cell profiles in patients stratified by cardiac diagnosis/imaging findings
Coagulation markers | Baseline
  Comparison of a panel of blood coagulation markers in patients stratified by cardiac diagnosis/imaging findings

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Tarkin, MBBS, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge Univeristy Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Corovic A, Zhao X, Huang Y, Newland SR, Gopalan D, Harrison J, Giakomidi D, Chen S, Yarkoni NS, Wall C, Peverelli M, Sriranjan R, Gallo A, Graves MJ, Sage A, Lyons PA, Sithole N, Bennett MR, Rudd JHF, Mallat Z, Zhao TX, Nus M, Tarkin JM. Coronavirus disease 2019-related myocardial injury is associated with immune dysregulation in symptomatic patients with cardiac magnetic resonance imaging abnormalities. Cardiovasc Res. 2024 Nov 25;120(14):1752-1767. doi: 10.1093/cvr/cvae159. PMID 39073768